CLINICAL TRIAL: NCT02268279
Title: A Phase 1, Open-label, Multi-center Study to Determine the Pharmacokinetics and Safety of Solithromycin as Add-on Therapy in Adolescents and Children With Suspected or Confirmed Bacterial Infection
Brief Title: Pharmacokinetics and Safety of Solithromycin in Adolescents and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE01-120
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Bacterial Infection
MeSH Terms: conditions — Bacterial Infections | interventions — solithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- solithromycin (Experimental): oral dosing (capsules and powder for suspension) by weight once per day intravenous dosing by weight once per day
  Interventions: Drug: solithromycin

INTERVENTIONS:
Drug: solithromycin
  Other Names: CEM-101

SUMMARY:
Pediatric study to evaluate the safety and pharmacokinetics of solithromycin (oral and intravenous) in children ages 0 to 17

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed bacterial infection with organisms against which solithromycin is expected to be active.

Exclusion Criteria:

* Serum creatinine >2 mg/dL
* Positive pregnancy test in females of childbearing potential
* History of intolerance or hypersensitivity to macrolide antibiotics

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2015-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of solithromycin in children and adolescents | 5 to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cohen-Wolkowiez, MD, Principal Investigator — Duke Clinical Research Institute
Locations (34):
- United States (31):
  - Little Rock, Arkansas
  - Orange, California
  - Palo Alto, California
  - San Diego, California
  - Jacksonville, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Iowa City, Iowa
  - Wichita, Kansas
  - Louisville, Kentucky
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - St Louis, Missouri
  - Omaha, Nebraska
  - Hackensack, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Brooklyn, New York
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Splendora, Texas
  - Richmond, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Bulgaria (3):
  - Plovdiv
  - Rousse
  - Sofia

REFERENCES:
- [Derived] Beechinor RJ, Cohen-Wolkowiez M, Jasion T, Hornik CP, Lang JE, Hernandez R, Gonzalez D. A Dried Blood Spot Analysis for Solithromycin in Adolescents, Children, and Infants: A Short Communication. Ther Drug Monit. 2019 Dec;41(6):761-765. doi: 10.1097/FTD.0000000000000670. PMID 31318840
- [Derived] Gonzalez D, James LP, Al-Uzri A, Bosheva M, Adler-Shohet FC, Mendley SR, Bradley JS, Espinosa C, Tsonkova E, Moffett K, Marquez L, Simonsen KA, Stoilov S, Boakye-Agyeman F, Jasion T, Hornik CP, Hernandez R, Benjamin DK Jr, Cohen-Wolkowiez M. Population Pharmacokinetics and Safety of Solithromycin following Intravenous and Oral Administration in Infants, Children, and Adolescents. Antimicrob Agents Chemother. 2018 Jul 27;62(8):e00692-18. doi: 10.1128/AAC.00692-18. Print 2018 Aug. PMID 29891609